CLINICAL TRIAL: NCT01084473
Title: Effect of Dexmedetomidine Infusion on Gastric Emptying and Gastrointestinal Transit in Healthy Volunteers
Brief Title: Effect of Dexmedetomidine on Gastric Emptying and Gastrointestinal Transit
Acronym: GADEX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Timo Iirola, Turku University Hospital and Turku University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: GADEX
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-03

CONDITIONS: Gastric Emptying; Healthy
Keywords: Dexmedetomidine; gastric emptying; oro-cecal transit time; Sedation in intensive care; Gastrointestinal effects of sedation
MeSH Terms: interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine (Experimental): The study subjects will be given a normal loading dose (1 μg/kg in 20 minutes) of dexmedetomidine (dexmedetomidine hydrochloride 100 μg/ml, Precedex® Abbott Laboratories North Chicago, IL 60064, USA) followed by continuous infusion of 0.7 μg/kg/h for 190 min. The administration of the loading dose will be started at t = -30 min (30 min prior to the administration of paracetamol and lactulose).
  Interventions: Drug: Dexmedetomidine
- Morphine (Active Comparator): The study subjects will be given 0.10 mg/kg morphine hydrochloride (morphine hydrochloride 2 mg/ml, Morphin® Nycomed Austria GmbH, St. Peter Strasse 25, A-4021, Linz, Austria) in 20 minutes followed by a placebo infusion for 190 min. The administration of the morphine infusion will be started at t = -30 min (30 min prior to the administration of paracetamol and lactulose).
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): The study subjects will be given a saline infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — The study subjects will be given a normal loading dose (1 μg/kg in 20 minutes) of dexmedetomidine (dexmedetomidine hydrochloride 100 μg/ml, Precedex® Abbott Laboratories North Chicago, IL 60064, USA) followed by continuous infusion of 0.7 μg/kg/h for 190 min. The administration of the loading dose will be started at t = -30 min (30 min prior to the administration of paracetamol and lactulose).
  Arms: Dexmedetomidine
Drug: Morphine — The study subjects will be given 0.10 mg/kg morphine hydrochloride (morphine hydrochloride 2 mg/ml, Morphin® Nycomed Austria GmbH, St. Peter Strasse 25, A-4021, Linz, Austria) in 20 minutes followed by a placebo infusion for 190 min. The administration of the morphine infusion will be started at t = -30 min (30 min prior to the administration of paracetamol and lactulose).
  Arms: Morphine
Drug: Placebo — 0.9 % NaCl will be infused.
  Arms: Placebo

SUMMARY:
The aim of the study is to determine the effect of dexmedetomidine infusion on gastric emptying and oro-caecal transit time in healthy volunteers, judged by measuring plasma paracetamol concentrations after paracetamol ingestion and pulmonary hydrogen measurement technique after lactulose ingestion. The effects of dexmedetomidine will be compared to the effects of morphine and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive function and fluent skills in the Finnish language in order to be able to give informed consent and communicate with the study personnel
* Age ≥ 18 years.
* Male gender.
* Weight ≥ 60 kg.
* Written informed consent from the subject.

Exclusion Criteria:

* Previous history of intolerance to the study drugs or related compounds and additives.
* Concomitant drug therapy of any kind except ibuprofen in the 14 days prior to the study days.
* Existing or recent significant disease.
* History of haematological, endocrine, metabolic or gastrointestinal disease.
* History of asthma or any kind of drug allergy.
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
* A positive test result for urine toxicology.
* A "yes" answer to any of the questions in a modified Finnish version of the Abuse Questions
* Donation of blood within six weeks prior to and during the study.
* Special diet or lifestyle factors which would compromise the conditions of the study or the interpretation of the results.
* BMI > 30 kg / m2.
* Participation in any other clinical study involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study.
* Smoking during one month before the start of the study or during the study period.
* Clinically significant abnormal findings in physical examination, ECG or laboratory screening [routine haematology (haemoglobin, haematocrit, red blood cell count, white blood cell count, platelets), renal function tests (creatinine, urea) and liver function tests (bilirubin)].

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The effect of dexmedetomidine on gastric emptying and oro-caecal transit time | 10, 15, 20, 30, 40, 45, 50, 60, 70, 75, 80, 90, 105, 120, 135, 150, 165, 180, 210 and 240 min
  5 ml venous blood samples will be collected immediately prior to administration of paracetamol (baseline) and thereafter at 10, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 135, 150, 165, 180, 210 and 240 min into EDTA tubes for determination of paracetamol plasma concentrations. End-expiratory breath samples will be obtained immediately prior to administration of lactulose (baseline) and thereafter at 15, 30, 45, 60, 75, 90, 105 and 120 min.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Iirola, MD, Principal Investigator — Turku University, Turku University Hospital
Locations (1):
- Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine, Turku University and Turku University Hospital, Turku, Finland